CLINICAL TRIAL: NCT01660178
Title: Profile of Newborn Undergoing Early Stimulation in a Neonatal Intensive Care Unit.
Status: Completed | Type: Observational
Sponsor: Universidade Federal do Rio de Janeiro (Other)
Responsible Party: Principal Investigator, karla camila lima de souza, camila souza, Universidade Federal do Rio de Janeiro
Other Study IDs: FDAAA
Record Dates: First submitted 2012-08-01; First posted 2012-08-08 (Estimated); Last update posted 2012-08-08 (Estimated); Status verified 2012-08

CONDITIONS: Motor Skills Disorders
Keywords: newborns; intensive care unit; early stimulation
MeSH Terms: conditions — Motor Skills Disorders

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To describe the profile of newborns undergoing early stimulation in a neonatal intensive care unit, characterizing the study population, according to its variables and neonatal risk factors, indications for treatment of early stimulation.

DETAILED DESCRIPTION:
Objective: To describe the profile of newborns undergoing early stimulation in a neonatal intensive care unit, characterizing the study population, according to its variables and neonatal risk factors, indications for treatment of early stimulation.

Methods: It was conducted a descriptive, cross-sectional and analytical study carried out in the General Hospital Dr. Cesar calls, from July to December 2010. The sample consisted of 116 medical records of newborns indicated for the treatment of early stimulation, representing (9.2%). The study excluded seven infants who had some type of congenital malformation. It was used the following variables: weight, sex, gestational age, Apgar score, diagnosis of Respiratory Distress Syndrome and Intracranial Hemorrhage and the use of mechanical ventilation and CPAP.

ELIGIBILITY:
Inclusion Criteria:

All cases of newborns who were admitted to the NICU and were referred for treatment of early stimulation

Exclusion Criteria:

all records relating to incomplete study variables and newborns who had a congenital malformation.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: newborns underwent early stimulation in a neonatal ICU
Sampling Method: Probability Sample
Dates: Start 2011-01; Study Completion 2011-06 (Actual)